CLINICAL TRIAL: NCT03569826
Title: Canadian Network for Autoimmune Liver Disease
Acronym: CaNAL
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CAPCR ID: 18-5951
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Primary Bilary Cirrhosis (PBC); Autoimmune Hepatitis; Overlap Syndrome
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Observational: There is no intervention being administered. This registry only observes patients through their regular standard of care visits.
  Interventions: Other: Observational; no intervention

INTERVENTIONS:
Other: Observational; no intervention — Observational; no intervention

SUMMARY:
CaNAL is a longitudinal observational cohort study of patients diagnosed with Primary Biliary Cholangitis (PBC), Autoimmune Hepatitis (AIH), or overlap syndrome. This study creates a nationwide registry and network focusing on high quality long-term follow-up of individual patient data from major Canadian centers.

Primary Biliary Cholangitis (PBC) and Autoimmune Hepatitis (AIH) are rare and slowly progressive liver diseases associated with development of cirrhosis, liver cancer (HCC) and liver failure requiring liver transplantation or leading to premature death. The rarity and slowly progressive nature of these autoimmune liver diseases make them difficult to study and only a large scale approach combining patient data from multiple centers across Canada will allow new insights. The primary aim of the Canadian Network for Autoimmune Liver Disease is to build a Canadian registry of patients with PBC, AIH, and overlap syndrome. We capture patient characteristics, laboratory assessments and natural history, patient-reported outcomes including quality of life measures and environmental exposures, response to treatment, and pre- and post-transplant outcomes. We will then identify risk factors associated with critical outcomes for the patient, including response to treatment, progression to transplant, risk of liver cancer, and recurrent disease after transplant. We can identify biomarkers (biochemical indicators of progression of disease) to help diagnose autoimmune liver disease at its earliest stages, ensuring timely treatment and preventing disease progression. CaNAL will provide a better understanding of autoimmune liver diseases, biomarkers predictive of disease progression or non-response to therapy as well as better knowledge of the etiology and pathogenesis. CaNAL will also help to serve as a platform for conducting clinical trials or targeted lab-studies to answer important questions that are unlikely to be evaluated by the pharmaceutical industry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Biliary Cholangitis and/or Autoimmune Hepatitis

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Primary Biliary Cholangitis and/or Autoimmune Hepatitis across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Liver transplant-free survival over time | Up to 6 years or time of death/liver transplant
  Time-to-event

SECONDARY OUTCOMES:
Biochemical values over time (e.g. aspartate aminotransferase, alkaline phosphatase, alanine aminotransferase, Bilirubin) | Through study completion, an average of 6 months
  Investigate trends of different biochemical values over time
Short Form 36 (SF-36) | Through study completion, an average of 6 months
  Health-Related Quality of Life
PBC-40 | Through study completion, an average of 6 months
  Health-Related Quality of Life, specific to Primary Biliary Cholangitis
5D Pruritus Scale | Through study completion, an average of 6 months
  Itch-Related Quality of Life through 5 dimensions: duration, degree, direction, disability, and distribution. Each dimension is scored from 1(lowest) to 5(highest) for a total score range of 5-25
Itch Visual Analog Scale | Through study completion, an average of 6 months
  Itch-Related Quality of Life; Continuous unitless itch scale from no itch to worst itch imaginable
Itch Numeric Rating Scale | Through study completion, an average of 6 months
  Itch-Related Quality of Life; Categorical integer scale from 0 (no itch) to 10 (worst itch imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hansen, PhD, Principal Investigator — University Health Network, Toronto General Hospital; Andrew Mason, MD, Principal Investigator — University of Alberta
Locations (15):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre (HDH Site), Kingston, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - McMaster University Medical Centre, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymized. A standardized electronic case record (e-CRF) form will be used to capture the data. The e-CRF form has been designed in REDCap, a secure web based application supporting data capture for research studies. REDCap is designed to comply with HIPAA security regulations. The CaNAL REDCap database (REDCap project CaNAL) has been established at the University of Alberta under the jurisdiction of the Women and Children's Health Research Institute (WCHRI).
  Individual centres will have access only to their own data and patient identifiers will only be visible to the individual centres. The steering committee will have access to all anonymized data within the REDCap database, that is without any patient identifiers. Main centres in Toronto and Edmonton will have access to de-identified data.
  Results will be disseminated via publication in international literature and presentation at international liver conferences. Patient data will be anonymous.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT03569826/Prot_SAP_000.pdf